CLINICAL TRIAL: NCT00239395
Title: A Randomised, Open-labelled Study to Compare the Efficacy and Safety of Meloxicam 7.5 mg IM Ampoules Once Daily and Meloxicam 7.5 mg Tablets Administered Orally Once Daily Over a Period of 7 Days in Patients With Osteoarthritis (OA)
Brief Title: A Study to Compare Meloxicam IM Once Daily and Meloxicam Administered Orally Once Daily in Patients With Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 107.265
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Meloxicam

INTERVENTIONS:
Drug: Meloxicam ampoule
Drug: Meloxicam tablet

SUMMARY:
The objective of this trial was to assess the efficacy and safety of 7.5 mg meloxicam i.m. once daily compared with 7.5 mg meloxicam tablets once daily p.o. in patients with osteoarthritis over a time period of 7 days.

DETAILED DESCRIPTION:
This was a randomized (1:1), open-label, multi-center, active-control, parallel-group study to compare the efficacy of 7.5 mg meloxicam i.m. once daily compared with 7.5 mg meloxicam tablets once daily p.o. in patients with osteoarthritis over a time period of 7 days.

The primary endpoint: Pain on active movement,

The secondary endpoint:

* Pain at rest
* Patient status with regard to change of arthritic condition assessed by the patient/investigator
* Patient's assessment of arthritic condition
* Onset of action
* Time to maximum pain relief
* Paracetamol consumption
* Withdrawals due to inadequate efficacy
* Final global assessment of efficacy by the patient/investigator

Safety endpoints

* Local tolerability assessment of the injections by the patient/investigator
* Patient's /Investigator's assessment of overall tolerability
* Number, nature and severity of adverse events
* Laboratory investigations
* Withdrawals due to safety reasons

Patients eligible for the trial who met all inclusion and exclusion criteria and who gave their informed consent were randomized to one of two treatment groups (i.e. meloxicam ampoule or meloxicam tablet).

The study period totaled 8-14 days included screening, randomisation, study drug administration, and 7-day follow-up. The relevant assessment were performed on the day of randomisation and 7-day follow up.

Study Hypothesis:

The null hypothesis of interest is that the primary endpoint for meloxicam ampoule is inferior to oral meloxicam. The alternative is that meloxicam ampoule is noninferior to the oral meloxicam .

Comparison(s):

The primary endpoint of the study was to assess pain on active movement by VAS prior and after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years or above
* Patients suffering from acute and painful exacerbation of osteoarthritis of the hip or knee.

The diagnosis must be based on

* clinical signs and symptoms or
* x-ray diagnosis plus clinical signs and symptoms

  * Assessment of pain on active movement (by the patient) must exceed 40 mm on a 100 mm visual analogue scale (VAS)
  * Symptoms of OA requiring administration of NSAIDs
  * Willingness and ability to provide written informed consent.

Exclusion Criteria:

* Known or suspected hypersensitivity to the trial drugs or their excipients, analgesics, antipyretics or NSAIDs
* Any clinical evidence of active peptic ulceration during the last six months
* Pregnancy or breastfeeding (precaution : attention should be drawn to reports that NSAIDs were reported to decrease the effectivity of intrauterine devices)
* Asthma, nasal polyps, angioneurotic oedema or urticaria following the administration of aspirin or NSAIDs
* Concomitant treatment with anti-coagulants (including heparin), lithium
* Concomitant administration of other NSAIDs or analgesic agents (except paracetamol up to 4g/day)
* Administration of any NSAID during the last 2 days (3 days for any oxicam) prior to the first administration of the trial drug
* Concomitant treatment with an oral corticosteroid initiated or with an altered dose over the previous month
* Parenteral or intraarticular administration of corticosteroids in the previous month
* Any i.m. injection during the previous 7 days
* Any contra-indication to i.m. injections
* Clinical evidence of or known severe cardiac, hepatic, renal, metabolic, haematological disease, mental disturbance, ulcerative colitis
* Any other rheumatological or non-rheumatological disease that could interfere with the evaluation of efficacy and safety
* Serum creatinine 125 % of the upper limit of normal range ; aspartate transferase (AST/SGOT) and/or alkaline transferase (ALT/SGPT) 200 % of the upper limit of normal range
* Platelet count < 100,000/mm3 ; leucocytes count < 3,000/mm3
* Synovectomy in the previous month or during the trial
* Participation in another clinical trial during this study or during the previous month
* Previous participation in this trial
* Patient unable to comply with the protocol
* Concomitant therapy with specific symptomatic drug of OA, such as chondroitin sulphate, diacerhein, initiated or with an altered dose over the previous 3 months.
* Intraarticular administration of hyaluronic acid in the previous month
* Patients where physiotherapy will be changed throughout the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168
Dates: Start 2004-07; Primary Completion 2004-12 (Actual); Study Completion 2004-12

PRIMARY OUTCOMES:
Pain on active movement by VAS. | day 0, day 7

SECONDARY OUTCOMES:
Pain at rest | up to 7 days
Patient status with regard to change of arthritic condition | up to 7 days
Withdrawals due to inadequate efficacy | up to 7 days
Onset of Analgesic action | up to 7 days
Time to maximum pain relief | up to 7 days
Paracetamol consumption | up to 7 days
Final global assessment of efficacy by patient | up to 7 days
Final global assessment of efficacy by investigator | up to 7 days
Assessment of local tolerability | up to 7 days
Nature and severity of adverse events | up to 7 days
Change in other laboratory investigations | up to 7 days
Withdrawals due to safety reasons | up to 7 days
Patient's and investigator's assessment of overall tolerability | up to 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim Shanghai
Locations (8):
- China (8):
  - People's Hospital, Beijing University, Beijing
  - Beijing Xuan Wu Hospital, Beijing
  - 1st Affiliated, Anhui Medical University, Hefei City, Anhui Province
  - Qilu Hospital, Shang Dong University, Nanzhou
  - Shanghai Renji Hospital, Shanghai
  - Shanghai Zhongshan Hospital, Shanghai
  - Shanghai Guanghai Hospital, Shanghai
  - Shanghai Changhai Hospital, Shanghai